CLINICAL TRIAL: NCT03636230
Title: Remote Patient Management of Cardiac Implantable Electronic Devices - Brady Devices
Brief Title: Remote Patient Management of CIEDs - Brady Devices
Acronym: RPM CIED Brady
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ratika Parkash (Other)
Collaborators: Cardiac Arrhythmia Network of Canada (Other); Medtronic (Industry); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Ratika Parkash, Staff Cardiologist Electrophysiologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-006
Record Dates: First submitted 2018-01-23; First posted 2018-08-17 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pacemaker
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Open label, 1:1 randomized trial, stratified by site and pacemaker dependence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Patient Management (Active Comparator): Remote monitoring only
  Interventions: Device: Remote Monitoring
- Standard of Care (Placebo Comparator): In-clinic visits
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Remote Monitoring — Remote Monitoring only + VIRTUES
  Arms: Remote Patient Management
Other: Standard of care — In-Clinic visits only
  Arms: Standard of Care

SUMMARY:
While remote monitoring (RM) technology is currently available and has permitted surveillance and device assessment from any patient location, the use has been inconsistent in Canada, where only 8500 out of a potential 120 000 patients with cardiac implantable electronic devices (CIEDs) are enrolled in this program. This technology is in widespread use worldwide for all CIEDs but in Canada, it is utilized primarily for implantable defibrillators, but not pacemakers. Whereas most of the trials were designed to evaluate the efficacy of RM in implantable cardioverter defibrillator (ICD) patients, in the pacemaker (PM) population, there has been work performed already to demonstrate an increase in detection of frequency of adverse clinical events and a reduction in reaction time to those events by RM. Based on all the available literature, it appears that RM benefits both patients and healthcare systems. Overall, studies have demonstrated that RM can be used safely in all device patient-populations, with the exception of pacemaker-dependent patients.

There have been no studies that have evaluated RM only follow up, nor have there been any studies evaluating pacemaker-dependent patients. This study that will safely assess the use of RM only, with in-clinic visits when necessary, that uses the patient-centered electronic platform developed by the Cardiac Arrhythmia Network of Canada (CANet) to perform PM follow up safely, in a more cost-effective manner.

DETAILED DESCRIPTION:
This is a Canadian multicenter randomized controlled trial to assess remote patient management. Patients will be randomized in a 1:1 fashion, stratified by pacemaker dependence and by center to either remote patient management of standard of care.

Remote patient management (intervention group):

* Patients will be followed by remote monitoring only. Transmissions will occur at six monthly intervals, with no in-clinic visits. If there is an actionable event on the remote transmission, patients will be seen at their closest community device clinic. The proposed intervention would eliminate any routine visits.
* Newly implanted pacemaker patients will be seen after the initial implant at the hub site, within 48 hours and then within 3 months to optimize programming for subsequent RM visits. Thereafter, all follow-up will occur through remote monitoring every six months. Unscheduled remote transmissions may also occur. Using a combination of remote monitoring, and novel technology, VIRTUES, patients will be managed outside of the clinic.
* Patients will be provided with real-time knowledge of success of their remote transmission and the status of the remote through a web-based portal called VIRTUES.
* Virtual patient record - all patient information in the intervention arm will be contained within an information cloud that will be accessible by patients; access to their own data may be granted by the patient themselves to permit delivery of care remotely, and to permit after hours follow up to be performed by the on call personnel.

Standard of care (comparison group):

The standard arm will be required to have in-clinic visits at yearly intervals. These patients would not have access to the virtual patient cloud or to remote monitoring.

Pacemaker programming: All patients in both arms will undergo programming as per the ASSERT II protocol (previously published) to optimize pacemaker parameters and detection of atrial and ventricular high rate episodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Medtronic or Abbott pacemaker capable of remote monitoring.
* Able to provide consent.
* Age >/= 18 years

Exclusion Criteria:

* No access to a family physician or general practioner
* Participation in the RPM CIED pilot study
* Unreliable automated capture verification function by the device in pacemaker-dependent patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 848 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to major adverse cardiac event (primary safety outcome) | 18 months
  Time to major adverse events (death, stroke, hospitalization for a cardiovascular cause, syncope or device-related emergency department visits). Survival free from the primary outcome will be estimated by the Kaplan-Meier method and compared, using the log-rank test. Cox proportional hazard regression analysis will be used to estimate the likelihood of survival, after verifying the proportional hazard assumption.
Cost effectiveness | 18 months
  Analysis will take the form of a cost utility analysis with cost effectiveness assessed in terms of the incremental cost per quality life year (QALY). Analysis will incorporate data on resource use and patient's utility values for the period from initiation of remote patient management to 12 months follow-up. Resource use associated with the remote patient management strategy will be estimated through detailed microcosting and will be contrasted with the costs of standard monitoring.
  QALYs will be estimated using the standard area under the cover methodology, controlling for baseline utility. Total costs and QALYs for each patient will be estimated with multiple imputation for missing data. The incremental costs and QALYs and incremental cost effectiveness ratios associated with remote patient management and the uncertainty around these will be derived through non-parametric bootstrapping.

SECONDARY OUTCOMES:
Quality of Life - Short Form (SF36) | 18 months
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health
Quality of Life - Florida Patient Acceptance Survey (FPAS) | 18 months
  The FPAS produces scores that range from 0-100, where higher scores indicate increased device acceptance.
Quality of Life - Florida Shock Anxiety Scale (FSAS) | 18 months
  The FSAS produces scores that range from 10-50. Higher scores signify increased shock anxiety.
Quality of Life - Brief Illness Perception Questionnaire (BIPQ) | 18 months
  Individual item analysis will be used in this study. The personal control score is the response to item 3. The treatment control score is the response to item 4. Illness concern is measured by item 6. This reflects a combination of emotional and cognitive representations. Scores on these individual items range from 0-10 where higher scores on personal and treatment concern are reflected in higher scores. Higher scores on illness concern are reflected in higher scores.
Device-related ER visits | 18 months
  Number of device-related ER visits (<24 hours)
Syncope | 18 months
  Rate of syncope
Time to detection of ventricular arrhythmia events | 18 months
  Any ventricular arrhythmia episodes detected by the pacemaker
Atrial fibrillation | 18 months
  AF detected by the pacemaker

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, MD FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (11):
- Canada (11):
  - Foothills Hospital, Calgary, Alberta
  - Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia
  - Memorial University of Newfoundland Hospital, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hopital Sacre Coeur, Montreal, Quebec
  - Hopital Laval, Québec, Quebec
  - Centre Hospitalier Universitaire du Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No